CLINICAL TRIAL: NCT03606148
Title: A Prospective Comparison of SurePathTM Liquid-based Cytology and Conventional Smear Cytology in Endoscopic Ultrasound-guided Sampling of Pancreatic Lesions
Brief Title: SurePathTM Liquid-based Cytology and Conventional Smear Cytology in Pancreatic Lesions
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 1803-094-930
Record Dates: First submitted 2018-04-26; First posted 2018-07-30 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2018-04

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SurePathTM: The subjects are randomly assigned to SurePathTM/Conventional test group at a ratio of 1: 1.
  In SurePathTM group, subjects who underwent SurePathTM liquid-phase cytology test with the first sample subjected to the conventional smear test with the second sample.
  Interventions: Diagnostic Test: SurePathTM
- Conventional: The subjects are randomly assigned to SurePathTM/Conventional test group at a ratio of 1: 1.
  In conventional test group, those who subjected to the conventional smear test with the first sample, will undergo the SurePathTM liquid cell test with the second obtained sample.
  Interventions: Diagnostic Test: SurePathTM

INTERVENTIONS:
Diagnostic Test: SurePathTM — In the liquid-phase cytology, a fine-aspirated sample is immediately inserted into a container containing a commercially available preservative solution without a separate slide-smearing procedure and immediately after the fine-needle aspiration.

SUMMARY:
The SurePathTM has been approved by the FDA since 1997. Currently, the SurePathTM is used for endometrial cells, body fluids, bronchoscopy aspirates, and thyroid fine needle aspirates. There is an advantage that the denaturation is small, the density of the cells is uniform, and the read area is small so that the read time can be shortened. Therefore, investigators plan to apply the SurePathTM test for pancreatic EUS-FNA specimens. Morphological comparative analysis is needed before completely replacing the existing classical smear test method. The aim of this study is to confirm that the SurePathTM is not inferior and is more accurate than the classical smear test.

ELIGIBILITY:
Inclusion Criteria:

* Patients who signed the agreement after the explanation
* Patients suspected of pancreatic cancer from radiological examinations (CT, MR, ultrasound)

Exclusion Criteria:

* Those who did not agree with the study
* Patients older than 18 years of age
* Serious mental patients
* Patients with severe accompanying diseases (ESRD, advanced COPD, severe heart failure, poorly controlled blood sugar)
* Pregnant women
* If EUS is difficult due to previous surgery (Billroth II or TG with R-en-Y)
* Patient with blood clotting abnormality
* If there is a risk of tract seeding after examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients above 18 years of age who underwent EUS-FNA for suspected pancreatic cancer based on imaging fingings.
Sampling Method: Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2018-04-17 (Actual); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy | 6 months after randomization
  If surgical treatment is performed after the examination, pathologic results of the surgical specimen and record will be checked whether it is malignancy or benign. If benign diagnosis is made by combining the results of SurePathTM and conventional smear test, the follow-up period is 6 months and the results of the 6-month follow-up imaging and additional biopsy are checked. Additional tests performed at this time are subject to the clinician's decision according to the clinical situation of each patient. The combined results make a final diagnosis and are compared between two groups.

SECONDARY OUTCOMES:
Sensitivity | 6 months after randomization
  The proportion of positives that are correctly identified as such.
Specificity | 6 months after randomization
  The proportion of negatives that are correctly identified as such

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Chun JW, Lee K, Lee SH, Kim H, You MS, Hwang YJ, Paik WH, Ryu JK, Kim YT. Comparison of liquid-based cytology with conventional smear cytology for EUS-guided FNA of solid pancreatic masses: a prospective randomized noninferiority study. Gastrointest Endosc. 2020 Apr;91(4):837-846.e1. doi: 10.1016/j.gie.2019.11.018. Epub 2019 Nov 20. PMID 31759036